CLINICAL TRIAL: NCT06201286
Title: Pain, Function and Range of Motion Related Outcomes of Mulligan Concept Applications in Obese Individuals With Chronic Mechanical Low Back Pain: a Randomized Controlled Study
Brief Title: Effect of Manual Therapy on Obese Individuals With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ömer Osman Pala, Assist. Prof, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AIBU-FTR-OOP-05
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Low Back Pain, Mechanical; Obesity
Keywords: Mulligan concept; Range of Motion; Low Back Pain; Obesity
MeSH Terms: conditions — Low Back Pain; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan group (MG) (Experimental): Mulligan group underwent an exercise program planned as 6 sessions. A one-day gap separated each session, and the entire program spanned 11 days. In Mulligan group, they received SNAG and NAGS techniques as part of the Mulligan concept applications, utilizing tools like the Mulligan belt, sponge, and stretcher. Both groups participated in supervised stretching and strengthening exercises.
  Interventions: Other: Mulligan Concept
- Control group (Other): Control group underwent an exercise program planned as 6 sessions. A one-day gap separated each session, and the entire program spanned 11 days. Both groups participated in supervised stretching and strengthening exercises.
  Interventions: Other: Stretching and strengthening exercises

INTERVENTIONS:
Other: Mulligan Concept — Mulligan Concept was applied by the physiotherapist who received A-B module trainings. Mulligan techniques were performed with 3 sets of 10 repetitions and 15-20 seconds rest between sets. Mobilisations were applied to the spinous process of each vertebra of the lumbar region with 3 sets of 10 repetitions of SNAG and 3 sets of 10 repetitions of NAGS techniques. In the standing position, the physiotherapist took a position next to the patient and stabilised the patient by grasping the abdomen with one arm.
  Strengthening exercises were applied to the rectus abdominis, internal and external obliquus, transversus abdominis muscles from flexor muscle groups in 3 sets of 10 repetitions. Stretching exercises were applied to the erector spinae and intertransversarii lumborum muscles from extensor muscle groups as 3 sets of 10 repetitions for 15-30 seconds.
  Arms: Mulligan group (MG)
Other: Stretching and strengthening exercises — Strengthening exercises were applied to the rectus abdominis, internal and external obliquus, transversus abdominis muscles from flexor muscle groups in 3 sets of 10 repetitions. Stretching exercises were applied to the erector spinae and intertransversarii lumborum muscles from extensor muscle groups as 3 sets of 10 repetitions for 15-30 seconds.
  Arms: Control group

SUMMARY:
This study will investigate the effectiveness of Mulligan mobilisation techniques Sustained Natural Apophyseal Glides (SNAGS) and Natural Apophyseal Glides (NAGs) on pain, disability, and range of motion (ROM) in obese individuals with mechanical low back pain (LBP).

DETAILED DESCRIPTION:
One of the most important methods in the treatment of LBP in recent years is manual therapy; manipulation, mobilisation and soft tissue techniques. With the manual techniques applied to the spine, the position and placement of the anatomical structures are changed and the tight and tense tissues are loosened. It has been observed that Mulligan techniques can correct the faults that cause pain in the spine and that the structures that cause pain return to their normal functions when released. In the literature, it has recently been observed that the number of studies examining manual therapy and Mulligan Concept methods has increased. Studies examining the effect of SNAG method on the lumbar region (12) and the effect of mobilisation and taping on chronic low back pain were found. However, no study was found in which SNAG and NAGS applications were applied on obese patients diagnosed with mechanical low back pain. Therefore, in this study, SNAG and NAGS in obese patients with LBP to investigate the effectiveness of the practices

ELIGIBILITY:
Inclusion Criteria:

diagnosed with mechanical low back pain, Body Mass Index (BMI) was between 30.00-39.99, 1.-2. Forty-six patients, aged 20-50 years, who were extremely obese and had pain radiating to the lower back and hips for at least 3 months,

Exclusion Criteria:

-

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | Two times in 11 day (before intervention, immediately after last intervention)
  Visual analogue scale (VAS) was used to assess the severity of mechanical neck pain. Individuals were asked to mark the pain they felt on a 10 cm long VAS scale ("0" indicates no pain and "10" indicates unbearable pain).
The Oswestry Low Back Pain Disability Questionnaire | Two times in 11 day (before intervention, immediately after last intervention)
  Evaluate back disability status a questionnaire consisting of 10 items. The items measure the severity of pain, self-care, lifting and carrying, walking, sitting, standing, sleeping, social life, travelling and the degree of change in pain, respectively. Under each item, the patient was asked six statements to be marked. The first statement is scored as "0" and the sixth statement is scored as "5". The higher the score, the higher the level of disability.
Joint Range of Motion Assessment (ROM) | Two times in 11 day (before intervention, immediately after last intervention)
  Active flexion, extension, right/left lateral flexion and rotation of the cervical region were measured in the sitting position with a phone goniometer application.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Osman PALA, PhD, Principal Investigator — Bolu Abant İzzet Baysal University
Locations (1):
- Faculty of Health Sciences Bolu Abant İzzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan for data sharing